CLINICAL TRIAL: NCT05100914
Title: A Nurse Empowered Spouses to Assist the Women With Breast Cancer Doing Daily Rehabilitation, and Evaluate the Effects on the Shoulder Range of Motion, Quality of Life, and Marital Intimacy.
Brief Title: Evaluation of the Effects of the Couple-based Family Nursing for Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Ting, Lin, Principal Investigator, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201900115B0
Record Dates: First submitted 2021-10-06; First posted 2021-10-29 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer; Women; Mastectomy; Breast-Conserving Surgery
Keywords: breast cancer; women; couple; family nursing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The Institute for Patient and Family-Centered Care promotes four core concepts: dignity and respect, information sharing, participation, and collaboration. Health care practitioners listen to and respect patients and families' perspectives and choices as well as incorporate the knowledge, values, beliefs, and cultural backgrounds of patients and families into the care plan. Affirmative and useful methods are employed for communicating data that are complete, accurate, and unbiased with patients and families, so that they receive data expediently, participate effectively, and make decisions in care. Health care practitioners encourage and support the families of patients for participation in caring and making decisions that align with families' preferences. Health care practitioners collaborate with patients and families in program development, implementation, and evaluation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The block randomization allocation sequence was computer-generated random numbers with a 1:1 ratio by Microsoft Excel. Participants were randomly allocated using sequentially numbered sealed envelopes. The envelopes were opened just before the operation, the research nurse who was involved in the data collection was blinded to the group allocation, and participants were not informed of their group allocation status. Given the nature of the interventions, it was not allowed to blind the participates and the research nurse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couple-based family nursing (Experimental): Women and their spouses were provided couple-based family nursing based on dignity and respect, information sharing, participation and collaboration for 30-60 minutes with couple-based interviews for arm rehabilitation. Arm rehabilitation begins within 48 hours postoperatively, and each movement should be incrementally increased in terms of exertion and repetition until the patient reaches 10 repetitions, 2-3 times daily, for one month.
  Interventions: Other: Couple-based family nursing
- Treatment as usual (Active Comparator): All women in the control group received hospital standard operative care, and couples attended a routine, 30-60-minute presentation about rehabilitation after breast surgery without any specific couple-based dyad interview.
  Interventions: Other: Couple-based family nursing

INTERVENTIONS:
Other: Couple-based family nursing — Spouses were taught the following rehabilitation movements: hand squeeze, wrist, and elbow flexion and extension, pendulum exercise, finger wall-climbing exercise, hair combing, wall pushup, pulley exercise, and turning around exercise. Arm rehabilitation begins within 48 hours postoperatively, and each movement should be incrementally increased in terms of exertion and repetition until the patient reaches 10 repetitions, 2-3 times daily, for one month. Spouses must support patients' wrist and elbow joints and maintain the arms perpendicular to the body. Spouses were instructed that if women experience negative emotions during the rehabilitation movements, spouses can express support to his wife through body language, such as kissing, holding hands, touching, or hugging.

SUMMARY:
The women with breast cancer and their spouses experienced physical and mental distresses together, nevertheless, the spouses were the significant supporters for patients during post-surgery rehabilitation. Based on the patient and family-centered care (PFCC), it was hypothesized that the couple engages in post-surgery rehabilitation could help women to have an improved shoulder range of movement, quality of life, and couples have better marital intimacy. All the women were eligible to be included in the randomized control trial if diagnosed with breast cancer, received breast surgery, her spouses were accompanying, and gave written consents. Women were randomized into two groups. The control group continues to receive usual care. The experimental group, who received couple-based family nursing (30-60 minutes couple-based interviews) based on the core concepts of PFCC: dignity and respect, information sharing, participation, and collaboration. The study nurse empowered spouses to assist the women's daily rehabilitation with a special workbook by clear pictures demonstration.

DETAILED DESCRIPTION:
Sample size: G*Power software was applied for estimating the sample size. Based on the relevant study "A couple-based intervention for female breast cancer" (Baucom et al., 2009), the median interpolated effect size across all female measures at posttest was 0.61. The type I error α was set at 0.05, statistical power was set at 0.8, and the effect size was set at 0.61 by using the independent sample t-test. We estimated a total sample number of 68, comprising the sample size of 34 for the experimental group and the sample size of 34 for the control group.

Method: The women with breast cancer and their spouses as couples were randomly allocated to the treatment as usual groups or couple-based family nursing groups in a 1:1 ratio by using computer-generated randomization. All eligible participants were recruited by a research assistant from the surgical wards. Participants were randomly allocated using sequentially numbered sealed envelopes. The envelopes were opened just before the operation, the research nurse who was involved in the data collection was blinded to the group allocation, and participants were not informed of their group allocation status. All participants were given a letter that contained the details of the research and informed the patients and spouses that they had the right to abstain from the research at any time, for any reason, and that participation and lack thereof would not affect their rights to treatment and care. Each participant was informed about the research and provided their written informed consent.

Couple-based family nursing: Besides the standard care and teaching program, the nurse researcher who has well trained about the breast cancer care family nursing and couple interviewing techniques. provided the women and their spouses a 30-60 minutes couple of interviews after the standard teaching program. The detail of the couple interview was followed the core concept of the Institute for Patient and Family-Centered Care (IPFCC, 2021), dignity and respect, information sharing, participation, and collaboration. The necessary caring knowledge was provided, the important value of couple together, and caring role to help their spouses to coach and help their wives to perform the rehabilitation during the critical hospitalization stage until to discharge back to home. In this intervention stage, the research nurse empowered their spouses to assist women with daily couple-based rehabilitation with a specific workbook that contained uncomplicated illustrations demonstrating what to expect during the first 48 hours after breast surgery. Firstly, we listened to couples' perspectives and assessed couples' knowledge and skills regarding arm rehabilitation; subsequently, we could understand spouses' willingness and values regarding assistance. Secondly, we provided comprehensive and unbiased data and clarified misinformation regarding arm rehabilitation. We taught couples the following rehabilitation movements: hand squeeze, wrist, and elbow flexion and extension, pendulum exercise, finger wall-climbing exercise, hair combing, wall pushup, pulley exercise, and turning around exercise. Arm rehabilitation begins within 48 hours postoperatively, and each movement should be incrementally increased in terms of exertion and repetition until the patient reaches 10 repetitions, 2-3 times daily, for one month. Spouses were required to support patients' wrist and elbow joints and maintain the arm perpendicular to the body. Spouses were instructed that if women experience negative emotions during the rehabilitation movements, spouses can express support to his wife through body language, such as kissing, holding hands, touching, or hugging. Thirdly, we investigated the concerns related to couples' practice rehabilitation movements. We explained to couples the distinctions between rehabilitation with and without spousal assistance to encourage couples to participate in this care program. Finally, we collaborated with each couple to develop an individualized rehabilitation program.

Data analysis: All data were analyzed using SPSS software version 24.0 and following intention-to-treat principles. Descriptive statistics of demographic and clinical characteristics were evaluated using chi-square tests for categorical variables. The outcome measures were analyzed at baseline and the group × time interaction effect between the two groups at one-month post-surgery by using a generalized estimating equation. The demographic and clinical characteristics were presented as numbers and percentages (%), the outcome measures were presented as means and standard deviations for participants. The level of significance was set at p < 0.05, and the intervention effects were considered to be significant at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage 0-3 breast cancer made by a specialist physician
* Women and spouses with a legal marriage
* Women and spouses aged ≥20 years
* Mastectomy or breast-conserving surgery
* Women and spouses with no history of mental illness
* Spouses who were willing to participate in postoperative care
* Women and spouses who could read and write in Chinese.

Exclusion Criteria:

* Women and spouses without a legal marriage
* Diagnosis of terminal breast cancer
* Women and spouses aged <20 years
* Planned or had undergone breast reconstruction
* Active chemotherapy or radiotherapy
* Women and spouses with a history of mental illness
* Women and spouses currently undergoing psychotherapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Shoulder range of motion | Change from Baseline Shoulder Range of Motion at one month
  The women's shoulder flexion, shoulder abduction, and shoulder external rotation, ranging from 0° to 180°.
Functional Assessment of Cancer Therapy-Breast | Change from Baseline Quality of Life at one months
  The quality of life of women with breast cancer, including physical well-being , social and family well-being , emotional well-being , functional well-being , and additional concerns-breast. The total score from 0 to 148, higher scores indicate more favorable quality of life of patients.
Marital intimacy inventory | Change from Baseline Marital Intimacy at one month
  The marital intimacy of couple, including spiritual intimacy , physical intimacy , sexual intimacy , social intimacy , and emotional intimacy. The total scores from 42 to 210, higher scores indicate more favorable marital intimacy.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chi Chiang, PhD, Study Chair — National Defense Medical Center
Locations (1):
- Yu-Ting Lin, Taipei, Neihu, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data were not approved by IRB.

REFERENCES:
- [Background] Andrzejczak E, Markocka-Maczka K, Lewandowski A. Partner relationships after mastectomy in women not offered breast reconstruction. Psychooncology. 2013 Jul;22(7):1653-7. doi: 10.1002/pon.3197. Epub 2012 Oct 9. PMID 23045167
- [Background] Baucom DH, Porter LS, Kirby JS, Gremore TM, Wiesenthal N, Aldridge W, Fredman SJ, Stanton SE, Scott JL, Halford KW, Keefe FJ. A couple-based intervention for female breast cancer. Psychooncology. 2009 Mar;18(3):276-83. doi: 10.1002/pon.1395. PMID 18702064
- [Background] Harris SR, Schmitz KH, Campbell KL, McNeely ML. Clinical practice guidelines for breast cancer rehabilitation: syntheses of guideline recommendations and qualitative appraisals. Cancer. 2012 Apr 15;118(8 Suppl):2312-24. doi: 10.1002/cncr.27461. PMID 22488705
- [Background] Ho PJ, Gernaat SAM, Hartman M, Verkooijen HM. Health-related quality of life in Asian patients with breast cancer: a systematic review. BMJ Open. 2018 Apr 20;8(4):e020512. doi: 10.1136/bmjopen-2017-020512. PMID 29678980
- [Background] Karki A, Simonen R, Malkia E, Selfe J. Postoperative education concerning the use of the upper limb, and exercise and treatment of the upper limb: cross-sectional survey of 105 breast cancer patients. Support Care Cancer. 2004 May;12(5):347-54. doi: 10.1007/s00520-004-0612-7. Epub 2004 Apr 3. PMID 15064932
- [Background] Kibar S, Dalyan Aras M, Unsal Delialioglu S. The risk factors and prevalence of upper extremity impairments and an analysis of effects of lymphoedema and other impairments on the quality of life of breast cancer patients. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12433. Epub 2016 Jan 13. PMID 26764197
- [Background] Levy EW, Pfalzer LA, Danoff J, Springer BA, McGarvey C, Shieh CY, Morehead-Gee A, Gerber LH, Stout NL. Predictors of functional shoulder recovery at 1 and 12 months after breast cancer surgery. Breast Cancer Res Treat. 2012 Jul;134(1):315-24. doi: 10.1007/s10549-012-2061-1. Epub 2012 Apr 19. PMID 22527107
- [Background] Li M, Chan CWH, Chow KM, Xiao J, Choi KC. A systematic review and meta-analysis of couple-based intervention on sexuality and the quality of life of cancer patients and their partners. Support Care Cancer. 2020 Apr;28(4):1607-1630. doi: 10.1007/s00520-019-05215-z. Epub 2019 Dec 24. PMID 31872299
- [Background] Li Q, Loke AY. A systematic review of spousal couple-based intervention studies for couples coping with cancer: direction for the development of interventions. Psychooncology. 2014 Jul;23(7):731-9. doi: 10.1002/pon.3535. Epub 2014 Apr 10. PMID 24723336
- [Background] Lopes VB, Lobo APA, Da Silva Junior GB, Melo AK, Lamboglia CG, Silva CABD. The experience of male spouses in the context of breast cancer: a systematic review of the literature. Psychol Health Med. 2018 Jan;23(1):89-98. doi: 10.1080/13548506.2017.1332374. Epub 2017 May 27. PMID 28552007
- [Background] Lovelace DL, McDaniel LR, Golden D. Long-Term Effects of Breast Cancer Surgery, Treatment, and Survivor Care. J Midwifery Womens Health. 2019 Nov;64(6):713-724. doi: 10.1111/jmwh.13012. Epub 2019 Jul 19. PMID 31322834
- [Background] Meleis AI, Sawyer LM, Im EO, Hilfinger Messias DK, Schumacher K. Experiencing transitions: an emerging middle-range theory. ANS Adv Nurs Sci. 2000 Sep;23(1):12-28. doi: 10.1097/00012272-200009000-00006. PMID 10970036
- [Background] McNeely ML, Binkley JM, Pusic AL, Campbell KL, Gabram S, Soballe PW. A prospective model of care for breast cancer rehabilitation: postoperative and postreconstructive issues. Cancer. 2012 Apr 15;118(8 Suppl):2226-36. doi: 10.1002/cncr.27468. PMID 22488697
- [Background] Ribeiro IL, Moreira RFC, Ferrari AV, Alburquerque-Sendin F, Camargo PR, Salvini TF. Effectiveness of early rehabilitation on range of motion, muscle strength and arm function after breast cancer surgery: a systematic review of randomized controlled trials. Clin Rehabil. 2019 Dec;33(12):1876-1886. doi: 10.1177/0269215519873026. Epub 2019 Sep 3. PMID 31480855
- [Background] Sharma A, Saneha C, Phligbua W. Effects of Dyadic Interventions on Quality of Life among Cancer Patients: An Integrative Review. Asia Pac J Oncol Nurs. 2021 Jan 29;8(2):115-131. doi: 10.4103/apjon.apjon_63_20. eCollection 2021 Mar-Apr. PMID 33688560
- [Background] Stefanut AM, Vintila M, Tudorel OI. The Relationship of Dyadic Coping With Emotional Functioning and Quality of the Relationship in Couples Facing Cancer-A Meta-Analysis. Front Psychol. 2021 Jan 8;11:594015. doi: 10.3389/fpsyg.2020.594015. eCollection 2020. PMID 33488460
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Wang F, Luo D, Fu L, Zhang H, Wu S, Zhang M, Zhou H, Sun T, Chen X. The Efficacy of Couple-Based Interventions on Health-Related Quality of Life in Cancer Patients and Their Spouses: A Meta-analysis of 12 Randomized Controlled Trials. Cancer Nurs. 2017 Jan/Feb;40(1):39-47. doi: 10.1097/NCC.0000000000000356. PMID 26925996
- [Background] Yang EJ, Park WB, Seo KS, Kim SW, Heo CY, Lim JY. Longitudinal change of treatment-related upper limb dysfunction and its impact on late dysfunction in breast cancer survivors: a prospective cohort study. J Surg Oncol. 2010 Jan 1;101(1):84-91. doi: 10.1002/jso.21435. PMID 19924721